CLINICAL TRIAL: NCT05300438
Title: A Multicenter, Open-label, Phase Ia/Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of TSN084 Tablets in Patients With Advanced Malignant Tumors.
Brief Title: Phase I Study of TSN084 in Patients With Advanced Malignant Tumors.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tyligand Bioscience (Shanghai) Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSN084-101US
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Cancer (With or Without Metastasis)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TSN084 (Experimental)
  Interventions: Drug: TSN084

INTERVENTIONS:
Drug: TSN084 — Oral tablets

SUMMARY:
TSN084 is a novel type II protein kinase inhibitor with demonstrated anti-tumor effects in vitro and in vivo and targets multiple tyrosine kinases, such as c-MET, FLT3, TRK and serine/threonine kinase CDK8/19. This first-in-human study is conducted to assess the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT), to evaluate the pharmacokinetics, safety and preliminary anti-tumor activity of TSN084 in advanced or metastatic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years old.
* The following three points are evaluated by the investigator and are deemed suitable to participate in the study: A. The subject fully understands the requirements of the study and voluntarily signs the written informed consent; B. Be able to comply with the medication requirements of the study and all study related procedures and evaluations; C. Not deemed as potentially unreliable and/or uncooperative.
* Meeting the requirements of tumor types shown below: Phase Ia Study: Histological or cytological diagnosis of locally advanced, relapsed, or metastatic malignancies, not amenable to standard therapy or for which no standard therapy is available. Phase Ib study: Histological or cytological diagnosis of the locally advanced, relapsed, or metastatic malignancies not amenable to standard therapy or for which no standard therapy is available. The specific tumor types/basket design with specific driven gene(s) will be determined by the principal investigator and the sponsor based on the Phase Ia study result.
* Survival expectations are ≥ 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 for Phase Ia, while 0 to 2 for Phase Ib. Subjects with advanced or metastatic malignancies who had at least one evaluable lesion during phase Ia study, while at least one measurable lesion during phase Ib study according to RECIST V1.1.
* Patients with adequate organ function at the time of screening (requiring no blood transfusion, no use of hematopoietic stimulating factor or human albumin within 14 days prior to screening), specifically defined as:

  1. Blood routine: Absolute neutrophil count (ANC) ≥ 1.5×109/L; Platelet count (PLT) ≥100×109/L; Hemoglobin (HGB) ≥ 90 g/L;
  2. Liver function: Serum Total bilirubin (TBIL) ≤ 1.5 Upper limit of normal value (ULN), and serum TBIL≤ 3×ULN in patients with liver metastasis or confirmed Gilbert syndrome. Alanine aminotransferase (ALT) and Aspartate transferase (AST) ≤ 2.5×ULN in subjects without liver metastasis; ALT or AST≤ 5×ULN in subjects with liver metastasis;
  3. Renal function: estimated creatinine clearance (CLcr) ≥ 60 mL/min as calculated using Cockcroft-Gault formula (Cockcroft DW 1976);
  4. Coagulation function: Activated Partial thromboplastin Time (APTT) and international normalized ratio (INR) ≤ 1.5×ULN (or within target range if on anticoagulation therapy);
  5. Cardiac function: Echocardiography (ECHO) shows left ventricular ejection fraction (LVEF) > 50%.
* Serum pregnancy test (for female of childbearing potential) negative within 3 days prior to first dosing of study treatment. Male and female patients of childbearing potential must agree to use effective methods of contraception from the time of first negative pregnancy test at screening, throughout the study and for 6 months after the last dose of the investigational product. A patient is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.

Exclusion Criteria:

* Has received any investigational agents within 21 days prior to the first administration of TSN084; or have stopped any investigational agents or other anti-tumors drugs for less than 5 half-lives or 21 days, whichever is longer;
* Acute toxic effects of prior anti-tumor therapy have not recovered to clinically significant NCI-CTCAE V5.0 grade ≤1 toxicity or baseline prior to the first administration of TSN084.
* At rest, the average Corrected QT interval (QTc, Fridericia's correction formula used) obtained by 12-lead Electrocardiograph (ECG) examination is > 470 ms (repeated 3 times). A variety of clinically significant arrhythmia, conduction, and resting ECG abnormalities, such as complete left bundle branch block, degree III, degree II, PR interval >250 ms. Various factors that may increase the risk of prolonged QTc or arrhythmia events, such as heart failure, hypokalemia, congenital long QT syndrome, a family history of long QT syndrome in a direct family member or sudden unexplained death before age 40, and use of any medications known to prolong QT intervals.
* Has an acute or chronic active hepatitis B defined as hepatitis B virus (HBV) DNA copy number ≥1×103 copies/mL or ≥ 200 IU/ml.
* Has acute or chronic active hepatitis C (HCV) defined as HCV-RNA level greater than the upper limit of the central reference value.
* Patients with active brain metastases will be allowed to enroll if their central nervous system (CNS) tumor metastases are confined to the supratentorial or cerebellum, have been adequately treated (surgery or radiotherapy), have maintained radiographic stability for at least 4 weeks, and do not require corticosteroids to control symptoms.
* Concurrent diseases that have not been controlled, such as:

  1. Severe infection, including but not limited to hospitalization due to infection, bacteremia, or severe pneumonia complications, occurs within 4 weeks prior to initiation of study treatment; Or patients who received therapeutic oral or intravenous antibiotics within two weeks prior to starting study treatment, and who received prophylactic antibiotics (e.g., for the prevention of urinary tract infection or chronic obstructive pulmonary disease);
  2. Symptomatic congestive heart failure (New York Heart Association Grades II-IV) or symptomatic or poorly controlled arrhythmias;
  3. Other malignancies (other than non-melanoma basal cell carcinoma or squamous cell carcinoma of the skin, breast/cervical carcinoma in situ, superficial bladder carcinoma that have received radical treatment and no evidence of disease recurrence) within 5 years prior to initiation of TSN084 treatment;
  4. Suspicion or confirmation of acute promyelocytic leukemia (for patients with acute myeloid leukemia) based on morphology, immune typing, molecular detection, or chromosome karyotype;
  5. Current subjects with cancerous meningitis, spinal cord compression, etc.;
  6. A history of poorly controlled hypertension;
  7. Symptomatic endogenous pulmonary disease;
  8. Any arterial thromboembolic event, including myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack, occurred within 6 months prior to enrolment;
  9. Significant malnutrition, such as the need for intravenous nutrient supplementation. Those who were stable for more than 4 weeks after correction of malnutrition before treatment of first dose of investigational product could be included.
  10. Tumor invasion of surrounding important organs or blood vessels (such as mediastinal great vessels, superior vena cava, trachea, esophagus, etc.), or at risk of esophagotracheal fistula or esophagopleural fistula;
  11. After endoesophageal or tracheal stent implantation;
  12. Other acute or chronic diseases or laboratory test abnormalities that may increase the risks associated with study participation or investigational product administration, or interfere with the interpretation of study results and, in the investigator's judgment, make subjects ineligible for study participation;
  13. Has a history of gastrointestinal perforation and/or fistula 6 months prior to the study enrollment;
  14. Uncontrolled third space effusion requiring repeated drainage, such as pleural effusion, ascites, pericardial effusion, etc. (Patients who do not need drainage effusion or have no significant increase in effusion after 3 days of cessation of drainage can be included).
* Expected to receive other anti-tumor therapies during the study (palliative radiotherapy is allowed).
* Allergic to TSN084 or its components.
* Has active gastrointestinal disease or other disease, or other factors such as surgical resection that may significantly affect drug absorption, metabolism, or excretion. This includes but not limited to the following conditions: malabsorption syndrome, inflammatory bowel disease, partial or complete intestinal obstruction, gastric or small intestinal resection.
* Has severe lung disease or history, such as moderate to severe chronic obstructive pulmonary disease (COPD), history of interstitial lung disease (ILD), drug-induced ILD, acute or chronic infectious pneumonia, lung transplantation, etc.
* Use of strong inducers or inhibitors of CYP3A drugs.
* Pregnant or lactating women.
* Dysphagia.
* Being involved in another interventional clinical study, or in an observational (non-interventional) clinical study, or in the follow-up phase of an interventional study.
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* Had a major surgical procedure (craniotomy, thoracotomy, laparotomy, vascular intervention, as defined by the investigator) within 4 weeks prior to the first administration of the investigational product, or had an unhealed wound, ulcer, or fracture. Note: For palliative care purposes, local surgical treatment of isolated lesions is acceptable.
* HIV infected patients (HIV 1/2 antibody positive).
* Known active syphilis infection, or active tuberculosis.
* Has a clear history of mental disorder with ongoing treatment.
* A history of drug abuse or drug use.
* The investigator believes that the subject may have other factors that may affect the results of the study and interfere with the subject's participation in the entire study process, including previous or existing physical conditions, abnormal treatment or laboratory tests, and the subject's unwillingness to comply with all procedures, restrictions and requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity | Every subject's DLT observation window is 28 days.
  Number of patients with dose limiting toxicity.
Incidence of Treatment-Emergent Adverse Events | From first dose to 28 ±7 days after last dose
  Incidence of adverse events, Treatment Emergent Adverse Event (TEAE), Serious Adverse Event (SAE), their relationship with the investigational product and respective severity. Adverse events and laboratory test values will be graded according to NCI-CTCAE V5.0.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | From first dose to day 1 in the second 28-day cycle
  To characterize the pharmacokinetic (PK) properties of TSN084 in patients with advanced malignant tumors.
Time to Cmax (Tmax) | From first dose to day 1 in the second 28-day cycle
  To characterize the pharmacokinetic (PK) properties of TSN084 in patients with advanced malignant tumors.
Area under the concentration versus time curve from time 0 to the last measurable concentration (AUC 0-t) | From first dose to day 1 in the second 28-day cycle
  To characterize the pharmacokinetic (PK) properties of TSN084 in patients with advanced malignant tumors.
Objective response rate (ORR) defined as the proportion of patients who have a CR or PR | From first dose to within 3 days of last dose.
  Tumor response assessments by the corresponding criteria by RECIST v1.1 to assess Objective response rate (ORR)
Duration of response (DoR) | From first dose to within 3 days of last dose.
  Tumor response assessments by the corresponding criteria by RECIST v1.1 to assess Duration of response (DoR).
Disease control rate (DCR) | From first dose to within 3 days of last dose.
  Tumor response assessments by the corresponding criteria by RECIST v1.1 to assess Disease control rate (DCR) after the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No